CLINICAL TRIAL: NCT05484401
Title: A Randomised, Double-blind, Double-dummy, Parallel-group, Single Dose, Active and Placebo-controlled Efficacy and Pharmacokinetics/Pharmacodynamics Study of 2 x 200 mg Ibuprofen Liquid Capsules for the Treatment of Pain After Surgical Removal of Impacted Third Molars.
Brief Title: Ibuprofen Liquid Capsules 2 x 200 mg Efficacy and PK/PD Study in Surgical Removal of Impacted Third Molars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5016401
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Tooth, Impacted; Tooth Diseases; Stomatognathic Diseases
Keywords: Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Non Narcotic; Analgesics
MeSH Terms: conditions — Tooth, Impacted; Tooth Diseases; Stomatognathic Diseases | interventions — Ibuprofen; Capsules; Tablets

STUDY DESIGN:
Intervention Model Description: The dental pain model used in this study is a robust and well established postsurgical pain model that produces pain that is predictable in its character, duration, and intensity. The model is widely accepted and has a proven record of assay sensitivity (i.e. separating active drugs from each other, as well as from placebo). The model is frequently used to evaluate NSAID type analgesics. Results from dental pain studies are accepted by the US Food and Drug Administration (FDA) and European authorities and have been widely extrapolated to other general pain conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, double dummy study. There will be two placebo tablets designed to be comparable to each of the active products (200mg Ibuprofen Liquid Capsules and 200mg Ibuprofen Tablets) in both shape, size, colour and weight. All subject packs have been designed and labelled to ensure blinding is maintained. Subjects, investigators and site staff will all be blind to the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Test Product (Experimental): Ibuprofen 200mg Oral Liquid Capsule, Placebo of Ibuprofen 200mg Oral Tablet
  Interventions: Drug: Ibuprofen 200Mg Oral Cap; Other: Placebo Tablets
- Reference Product (Active Comparator): Ibuprofen 200mg Oral Tablet, Placebo of Ibuprofen 200mg Oral Liquid Capsule
  Interventions: Drug: Ibuprofen 200Mg Oral Tablet; Other: Placebo Liquid Capsule
- Placebo (Placebo Comparator): Placebo of Ibuprofen 200mg Oral Liquid Capsule, Placebo of Ibuprofen 200mg Oral Tablet
  Interventions: Other: Placebo Liquid Capsule; Other: Placebo Tablets

INTERVENTIONS:
Drug: Ibuprofen 200Mg Oral Cap — 2 x 200mg Liquid Capsules once in 12 hours
  Other Names: Test Product; 200mg Ibuprofen Liquid Capsule; Nurofen 200mg Ibuprofen Liquid Capsule
  Arms: Test Product
Drug: Ibuprofen 200Mg Oral Tablet — 2 x 200mg Tablets once in 12 hours
  Other Names: Reference Product; 200mg Ibuprofen Tablet; Nurofen 200mg Ibuprofen Tablet
  Arms: Reference Product
Other: Placebo Liquid Capsule — 2 x Liquid Capsules once in 12 hours
  Arms: Placebo; Reference Product
Other: Placebo Tablets — 2 x Tablets once in 12 hours
  Arms: Placebo; Test Product

SUMMARY:
This is a single centre, three-arm randomised, double-blind, double-dummy, parallel group, single-dose, active and placebo-controlled efficacy and pharmacokinetics/ pharmacodynamics study to evaluate the efficacy and safety of 2 x 200 mg Ibuprofen Liquid Capsules in subjects with post-operative dental pain.

DETAILED DESCRIPTION:
Eligible subjects will complete all screening procedures within 28 days before the surgery and randomisation.

At Screening, subjects will provide written informed consent to participate in the study before any protocol specified procedures or assessments are completed. On Day 1, subjects who continue to be eligible for study participation after completing screening procedures and assessments will undergo extraction of 2 or more third molars. At least 1 of the third molars must be a fully or partially bone impacted mandibular molar.

All subjects will receive local anaesthesia (2% lidocaine with 1:100,000 epinephrine). Nitrous oxide will be allowed at the discretion of the investigator. Subjects who experience moderate to severe pain intensity (a score of ≥ 5 on a numeric rating scale [NRS] from 0-10 where 0 = no pain, 10 = worst pain ever) within 6 hours after surgery and who continue to meet all study entry criteria will be randomised in a 3:3:1 ratio to receive a single dose of 2×200 mg Ibuprofen Liquid Capsules, 2×200 mg ibuprofen tablets, or placebo. The randomisation will be stratified by baseline pain category (moderate or severe) using a categorical scale based on the NRS score that includes the categories of none (0), mild (1-4), moderate (5-7), and severe (8-10).

Subjects will re-assess their baseline pain intensity using the NRS immediately before receiving study drug (pre-dose, Time 0) and their pain intensity (NRS) and pain relief (5 point categorical scale) at the following time points (pre-dose, 10, 20, 30 and 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours after Time 0; and immediately before each dose of rescue medication, if any. For assessments less than 1 hour apart a window of +/-2 min is allowable whilst for assessments at least 1 hour apart a +/-5 min window is allowable.

The double stopwatch method will be used to record the time to perceptible pain relief and time to meaningful pain relief during the 8 hours following the first dose or until subject takes rescue medication. Subjects will complete a global evaluation of study drug and satisfaction with pain relied assessment 12 hours (+/- 5 minutes) after Time 0 or immediately before the first dose of rescue medication (whichever occurs first). Vital signs will be recorded after the subject has been in a sitting position for 3 minutes at the following times: before surgery, within 30 minutes before Time 0, 12 hours after Time 0, immediately before the first dose of rescue medication(if required) and at the follow-up visit. Adverse events (AEs) will be monitored and recorded from the time of signing of the informed consent form (ICF) until the Follow up Visit (or Early Termination Visit). During the 12 hours following Time 0, subjects will complete efficacy and safety assessments. Subjects will remain at the study site overnight and will be discharged on Day 2.

Paracetamol / acetaminophen (1000 mg) will be permitted as the initial rescue medication. Subjects will be encouraged to wait at least 60 minutes after receiving study drug before taking rescue medication. If acetaminophen rescue medication is not effective in relieving the subject's pain, 5 mg oxycodone rescue medication may be administered at the discretion of the investigator.

Subjects are not permitted to take any concomitant medications that might confound assessments of pain relief, such as psychotropic drugs, antidepressants, sedative-hypnotics (other than those permitted for conscious sedation), or other analgesics taken within five times of their elimination half-lives (other than those used at the surgery).

Other restrictions include the following: alcohol use is prohibited from 24 hours before surgery until discharge on Day 2; Food will be restricted from midnight before surgery until 4 hour after surgery; during this time, water may be permitted up to 2 hours prior to surgery and a single drink of 8 fluid ounces of water with their treatment, water will not be permitted until 1 hour post dose. Vaccinations should not have been administered 7 days prior to surgery, subjects should avoid strenuous physical activity from 72 hours prior to dosing, and will not be permitted to smoke or use nicotine containing products for the duration of their involvement in the study.

A subset of 70 subjects will be randomly selected from the study population to take part in a Pharmacokinetic sub study. Blood samples will be collected at 10, 15, 20, 30 and 45 minutes and 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post dose.

Upon discharge from the study site, subjects may be prescribed pain medication for use at home according to the standard practice of the study site. On Day 8 (± 2 days), subjects will return to the study site for an abbreviated confirmatory physical assessment and AE assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent (for subjects who are below the age of legal consent, parent(s) or legally authorized representative(s) provides written informed consent and the subject provides written assent).
* Subject is male or female and aged ≥16 and ≤55 years of age at screening.
* Requires extraction of 2 or more third molars. At least 1 of the third molars must be a fully or partially bone impacted mandibular molar.
* Experiences moderate to severe pain intensity within 6 hours after surgery, as measured by a NRS score of ≥ 5 on a 0-10 scale.
* Has a body weight ≥ 45 kg and a BMI ≥17 kg/m2 and ≤ 30 kg/m2.
* Female subjects or the female partners of male subjects of childbearing potential must be using a highly effective method of contraception for at least one month prior to screening, throughout the study and for one menstrual cycle after last drug administration. [A highly effective method of contraception is defined as a method that can achieve a low failure rate of less than 1% per year when used consistently and correctly. Such methods include combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, injectable & implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomised partner (who has received medical assessment of the surgical success), or sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments and must be the preferred and usual lifestyle of the subject)].
* Free of clinically significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
* Is willing and able to comply with study requirements (including diet and smoking restrictions), complete the pain evaluations, remain at the study site overnight (if necessary) and return for follow-up 7 (± 2) days after surgery, (Day 8 ± 2 days).

Exclusion Criteria:

* Known hypersensitivity reactions or allergy (e.g. asthma, rhinitis, angioedema or urticaria) in response to nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen), acetylsalicylic acid (aspirin), ingredients of the study drug, or any other drugs used in the study, including anaesthetics and antibiotics that may be required on the day of surgery.
* In the opinion of the investigator, any subject with a clinically relevant history of peptic ulceration, gastrointestinal bleeding or perforation, heart failure, renal or hepatic failure, uncontrolled hypertension, nasal polyps, or chronic rhinitis.
* In the opinion of the investigator, the participant has a clinically significant history of asthma or a documented intolerance to NSAIDs resulting in exacerbation of symptoms.
* Has complications from the tooth extraction or any other clinically significant medical history that, in the opinion of the investigator, would affect the subject's ability to comply or otherwise contraindicate study participation, including but not limited to the following: cardiac, respiratory, gastroenterological, neurological, psychological, immunological, haematological, oncological, or renal disease.
* Has undergone another dental surgery within 60 days prior to the day of surgery.
* A positive urine drugs of abuse test at screening and during the study (with the exception of a positive drugs of abuse screen that is a consequence of permitted prescription medicines) or positive alcohol breathalyser test during the study.
* If female, has a positive pregnancy test at screening (serum) or on the day of surgery prior to surgery (urine), or is lactating.
* Has known or suspected, (in the opinion of the investigator), history of alcoholism or drug abuse within 2 years of screening or evidence of tolerance or physical dependence before dosing with study drug.
* Is a current smoker (including any nicotine products e.g., e-cigarettes or chewing tobacco) or ex-smoker who has smoked or used nicotine replacement products within 1 year of screening
* Taking any concomitant medications that might confound assessments of pain relief, such as psychotropic drugs, antidepressants, sedative-hypnotics (other than those permitted for conscious sedation), or other analgesics taken within five times of their elimination half-lives.
* Those taking medicinal products prone to drug-drug interactions described in the investigator's brochure [IB]. These include Acetyl Salicylic Acid, other NSAIDs including cyclo-oxygenase-2 selective inhibitors, anticoagulants, antihypertensives (ACE inhibitors and Angiotensin II receptor antagonists) and diuretics, corticosteroids, anti-platelet agents and Selective Serotonin Re-uptake Inhibitors (SSRIs), cardiac glycosides, lithium, methotrexate, ciclosporin, mifepristone, tacrolimus, zidovudine and quinolone antibiotics.
* Is considered by the investigator, for any reason (including, but not limited to the risks described as precautions, warnings and contraindications in the current version of the investigator's brochure [IB] for 200 mg ibuprofen liquid capsules), to be an unsuitable candidate to receive the study drug.
* Has a history of chronic use (defined as daily use for > 2 weeks) of nonsteroidal anti-inflammatory (NSAIDs, including topical), opiates, or corticosteroids (except inhaled nasal steroids), for any condition within 3 months before dosing with study drug.
* Has significant difficulties swallowing capsules or tablets or is unable to tolerate oral medication.
* Subject has received an investigational product or participated in another trial involving a marketed or investigational drug in the 90 days (or for investigational agents with a long half-life, a washout of 5 half-lives) prior to first drug administration (washout period between studies is defined as the period of time elapsed between the last dose of the previous study and first dose for this study). Or if the investigator believes that any previous participation in an investigational study would be to the detriment of the safety of the participant or the conduct of the study.
* Enrolment of the Investigator, his/her family members, employees and other dependent persons.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 294 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference 0-8 hours (SPID0-8) vs placebo using the Numeric Rating Scale (NRS) for pain | 0-8 hours
  SPID0-8 will be used to compare the test product against the placebo product. Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 8 hour timepoint, the SPID0-8 will be take as the area under the curve. The NRS will be used to assess the Pain Intensity, the NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Time to Meaningful pain relief vs active comparator using double stopwatch method | 0-8 hours
  Time to onset of meaningful pain relief (measured as time to meaningful pain relief) using double stopwatch will be used to compare the test product with the active comparator. Two stopwatches will be started immediately after the subject has swallowed the study drug with 8 ounces of water. Each subject will be instructed, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). The subject will also be instructed, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). If the subject does not press the stopwatches within 8 hours after Time 0 the subject will discontinue use of the stopwatches.

SECONDARY OUTCOMES:
Time to onset of pain relief using double stopwatch method vs Placebo | 0-8 hours
  Time to onset of meaningful pain relief (measured as time to perceptible pain relief confirmed by time to meaningful pain relief) using double stopwatch will be used to compare test product with placebo. Two stopwatches will be started immediately after the subject has swallowed the study drug with 8 ounces of water. Each subject will be instructed, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). The subject will also be instructed, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). If the subject does not press the stopwatches within 8 hours after Time 0 the subject will discontinue use of the stopwatches.
Total Pain Relief 0-6 hours (TOTPAR6) for Test Product vs Active Comparator After Time 0 | 0-6 hours
  TOTPAR6 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to active comparator. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 6 hour timepoint, TOTPAR6 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Proportion of subjects using rescue medication vs Active Comparator | 0- 6 hours
  Proportion of subjects using rescue medication within the first 6 hours will be used to compare the test product against active comparator
Time to first use of rescue medication vs Active Comparator | 0-12 hours
  Time to first use of rescue medication will be used to compare the test product and active comparator.
Time to onset of pain relief using double stopwatch method vs Active Comparator | 0-8 hours
  Time to onset of meaningful pain relief (measured as time to perceptible pain relief confirmed by time to meaningful pain relief) using double stopwatch will be used to compare test product with Active Comparator. Two stopwatches will be started immediately after the subject has swallowed the study drug with 8 ounces of water. Each subject will be instructed, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). The subject will also be instructed, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). If the subject does not press the stopwatches within 8 hours after Time 0 the subject will discontinue use of the stopwatches.
Proportion of Subjects achieving at least "a lot" of pain relief at 1 and 2 hours post dose vs Placebo and Active Comparator | 0-2 hours
  Proportion of subjects achieving at least "a lot" of pain relief measured using PRS at 1 and 2 hours after Time 0 will be used to compare the test product (2 x 200 mg Ibuprofen Liquid Capsules) against active comparator (2 x 200 mg standard ibuprofen tablets) and the test product (2 x 200 mg Ibuprofen Liquid Capsules) against placebo. The PRS will be used to measure pain relief and is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Proportion of subjects using rescue medication vs Placebo | 0-6 hours
  Proportion of subjects using rescue medication within the first 6 hours will be used to compare the test product against Placebo
Proportion of subjects using rescue medication vs Placebo and Active Comparator | 0-12 hours
  Proportion of subjects using rescue medication within the first 12 hours will be used to compare the test product against Placebo and Active Comparator
Time to peak pain relief using Pain Relief Scale (PRS) vs active comparator and placebo | 0-12 hours
  The time to reach peak pain relief will be compared vs active comparator and placebo. The PRS will be used to measure pain relief and is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Proportion of subjects with "Complete" pain relief at 30 minutes, assessed using PRS, after Time 0 vs Active Comparator and Placebo | 0-12 hours
  The proportion of subjects with complete pain relief at 30 minutes, assessed using PRS after T 0 will be compared vs active comparator and placebo. The PRS will be used to measure pain relief and is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Proportion of subjects with "Complete" pain relief at 30 minutes, assessed using PRS, after Time 0 vs Active Comparator and Placebo | 0-30 minutes
  The proportion of subjects with at least a 50% decrease in pain intensity at 30 minutes after T0 (using NRS for pain) compared to active comparator and placebo. The NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Proportion of subjects with at least 50% decrease in pain intensity at any time 6 hours after T0 using NRS vs active comparator and placebo | 0-6 hours
  The proportion of subjects with at least a 50% decrease in pain intensity at any time 6 hours after T0 (using NRS for pain) compared to active comparator and placebo. The NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Time to first use of rescue medication vs Placebo | 0-12 hours
  Time to first use of rescue medication will be used to compare the test product and placebo.
Total Pain Relief 0-2 hours (TOTPAR2) for Test Product vs Active Comparator After Time 0 | 0-2 hours
  TOTPAR2 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to active comparator. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 2 hour timepoint, TOTPAR2 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Total Pain Relief 0-4 hours (TOTPAR4) for Test Product vs Active Comparator After Time 0 | 0-4 hours
  TOTPAR4 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to active comparator. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 4 hour timepoint, TOTPAR4 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Total Pain Relief 0-8 hours (TOTPAR8) for Test Product vs Active Comparator After Time 0 | 0-8 hours
  TOTPAR8 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to active comparator. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 8 hour timepoint, TOTPAR8 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
PK Subset: Cmax will be evaluate for each treatment (test and active comparator) | 0-12 hours
  The Cmax (Maximum Plasma Concentration) will be calculated for the test and active comparator.
PK Subset: tmax will be evaluate for each treatment (test and active comparator) | 0-12 hours
  The tmax (Time of maximum plasma concentration) will be calculated for the test and active comparator.
PK Subset: AUC0-t will be evaluate for each treatment (test and active comparator) | 0-12 hours
  The AUC0-t (Area under the plasma concentration-time curve from time zero to the last quantifiable plasma concentration) will be calculated for the test and active comparator.
PK Subset: tlag will be evaluate for each treatment (test and active comparator) | 0-12 hours
  The tlag (the time delay between drug administration and first observed concentration) will be calculated for the test and active comparator.
Minimum Effective Concentration (MEC) for onset of analgesia (SC1) and meaningful pain relief (SC2)- test product (TP) and active comparator (AC), and combined (COM) | 10-90mins
  The proportion of subjects with confirmed pain relief (assessed via timepoint 1 in the double stopwatch method) at 10, 15, 20, 30, 45, 60, 75 and 90 minutes. The first timepoint at which the incidence of confirmed time to onset of pain (stop clock 1, SC1) is statistically significantly (p<0.05) greater than placebo will be calculated for each treatment group, these will be termed SC1(TP) for the test product and SC1(AC) for the active comparator. The same methodology will be followed to determine the first timepoint at which the confirmed meaningful pain relief (timepoint 2 in the double stopwatch method) at 10, 15, 20, 30, 45, 60, 75 and 90 minutes is statistically significantly greater (p<0.05) than placebo will be calculated for each treatment group, these will be termed SC2(TP) and SC2(AC). The mean ibuprofen plasma concentration (including chiral analysis) by treatment group (and combined) is considered the minimum effective concentration.
Occupancy Time | 0-12 hours
  Occupancy time will be calculated for both test and comparator products individually and as a combination, a ratio of time where ibuprofen (both racemic and s enantiomer) plasma levels are above MEC.SC1 and MEC.SC2 will be reported for the test product, active comparator and a combination of the two.
Time to meaningful pain relief compared to the placebo | 0-8 hours
  Time to onset of meaningful pain relief (measured as time to perceptible pain relief confirmed by time to meaningful pain relief) using double stopwatch will be used to compare the test product with the placebo. Two stopwatches will be started immediately after the subject has swallowed the study drug with 8 ounces of water. Each subject will be instructed, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). The subject will also be instructed, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). If the subject does not press the stopwatches within 8 hours after Time 0 the subject will discontinue use of the stopwatches.
Total Pain Relief 0-2 hours (TOTPAR2) for Test Product vs Placebo | 0-2 hours
  TOTPAR2 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to Placebo. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 2 hour timepoint, TOTPAR2 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Total Pain Relief 0-4 hours (TOTPAR4) for Test Product vs Placebo | 0-4 hours
  TOTPAR4 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to Placebo. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 4 hour timepoint, TOTPAR4 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Total Pain Relief 0-6 hours (TOTPAR6) for Test Product vs Placebo | 0-6 hours
  TOTPAR6 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to Placebo. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 6 hour timepoint, TOTPAR6 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Total Pain Relief 0-8 hours (TOTPAR8) for Test Product vs Placebo | 0-8 hours
  TOTPAR8 after Time 0 will be assessed using the Pain Relief Scale (PRS) will be used to compare test product to Placebo. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 8 hour timepoint, TOTPAR4 is the area under the curve. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Pain intensity Score at each scheduled timepoint After Time 0 | 0-12 hours
  Pain intensity score at each scheduled time point will be assessed using a numeric rating scale (NRS) for pain. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain
Pain intensity difference score at each scheduled timepoint after Time 0. | 0-12 hours
  Pain intensity score at each scheduled time point will be assessed using a numeric rating scale (NRS) for pain. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain
Summed Pain Intensity Difference over 0 to 2 hours (SPID2), test product vs active comparator and test vs against placebo using the Numeric Rating Scale (NRS) for pain. | 0-2 hours
  SPID2 will be used to compare the test product against the comparator and placebo product. Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 2 hour timepoint, the SPID2 will be take as the area under the curve. The NRS will be used to assess the Pain Intensity, the NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Summed Pain Intensity Difference over 0 to 4 hours (SPID4), test product vs active comparator and test vs against placebo using the Numeric Rating Scale (NRS) for pain. | 0-4 hours
  SPID4 will be used to compare the test product against the comparator and placebo product. Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 4 hour timepoint, the SPID4 will be take as the area under the curve. The NRS will be used to assess the Pain Intensity, the NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Summed Pain Intensity Difference over 0 to 6 hours (SPID6), test product vs active comparator and test vs against placebo using the Numeric Rating Scale (NRS) for pain | 0-6 hours
  SPID6 will be used to compare the test product against the comparator and placebo product. Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 2 hour timepoint, the SPID0-2 will be take as the area under the curve. The NRS will be used to assess the Pain Intensity, the NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain.
Time to first perceptible pain relief. | 0-8 hours
  Two stopwatches were started immediately after the subject swallowed the study drug. Subjects were instructed to, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). Time to first perceptible pain relief was date/time of the first reported pain relief (any) as assessed by the subject (i.e., when the subject stopped the first stopwatch, irrespective of the second) - date/time of the first dose of study drug. If the stopwatch were not stopped within 8 hours after Time 0, use of the stopwatches was discontinued.
Pain relief score at each scheduled time point after Time 0. | 0-12 hours
  Pain relief score at each scheduled time point after Time 0 was measured using the Pain Relief Scale (PRS). The PRS was used to measure pain relief and is a 5-point categorical scale, with response choices of: none = 0; a little = 1; some = 2; a lot = 3; and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome.
Subject's global evaluation of study drug. | 0-12 hours
  Patient's global evaluation of study drug using 5 point categorical scale, response choices of 0 = poor, 1 = fair, 2 = good, 3 = very good, or 4 = excellent to be completed by the patient in response to the question "How effective do you think the study drug is as a treatment for pain?". Subjects will complete the global evaluation of study drug 24 hours after Time 0 or immediately before the first dose of rescue medication (whichever occurs first).
Subject satisfaction with pain relief. | 0-12 hours
  Patient's global evaluation of pain relief using 5 point categorical scale, response choices of Very Satisfied, Satisfied, Neither Satisfied nor Dissatisfied, Dissatisfied or Very Dissatisfied to be completed by the patient in response to the question "How satisfied are you with the pain relief provided by the study medication?". Subjects will complete the global evaluation of study drug 24 hours after Time 0 or immediately before the first dose of rescue medication (whichever occurs first).
Peak pain relief. | 0-12 hours
  Peak pain relief at each time point will be measured using the Pain Relief Scale (PRS). The PRS will be used to measure pain relief and is a 5-point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. The peak pain relief each subject achieved will be summarised.
Summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 4 hours (SPRID4). | 0-4 hours
  Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 4 hour timepoint, the SPID4 will be calculated as the area under the curve. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 4 hour timepoint, TOTPAR4 is the area under the curve. SPRID4 is SPID4 + TOTPAR4. The PRS was used to measure pain relief and is a 5-point categorical scale with response choices of: none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. An 11-point (0-1) NRS for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain.
Summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 8 hours (SPRID8). | 0-8 hours
  Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 4 hour timepoint, the SPID8 will be calculated as the area under the curve. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 8 hour timepoint, TOTPAR8 is the area under the curve. SPRID8 is SPID8 + TOTPAR8. The PRS was used to measure pain relief and is a 5-point categorical scale with response choices of: none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. An 11-point (0-1) NRS for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain.
The summed pain intensity difference (SPID) over 0 to 8 hours (SPID8) will be used to compare the test product and active comparator product. | 0-8 hours
  SPID8 was used to compare the test product to the comparator product. Pain Intensity Difference (Difference in NRS for baseline and each timepoint) will be plotted against timepoint up to the 8 hour timepoint, the SPID0-8 will be take as the area under the curve. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain.
Proportion of subjects who achieve at least 50% of the maximum TOTPAR (maxTOTPAR) over 0 to 6 hours will be used to compare the test product against active comparator and the placebo | 0-6 hours
  The proportion of subjects who achieve at least 50% of the maxTOTPAR in the first 6 hours will be used to compare the test product to comparator and placebo test groups. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 6 hour timepoint, TOTPAR6 is the area under the curve. The maxTOTPAR is the maximum total pain relief score (TOTPAR) possible up to and including the 6 hour timepoint. Each subjects TOTPAR will be assessed against the maxTOTPAR and the proportion who reach a value of at least 50% of this value will be used to assess this endpoint. The Pain Relief Scale (PRS) will be used to measure pain relief and is a 5-point categorical scale with response choices of: none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome.
Relationship between speed of onset of pain relief and overall pain over 0-60 minutes. | 0-1 hours
  To assess the relationship between speed of onset of pain relief and overall pain experience by evaluating the association between the slope of the change in pain intensity over 0-60 minutes and %maxTOTPAR over 0-60 minutes. Pain Intensity scores using the NRS will be plotted against each timepoint up to the 1 hour timepoint. Pain Relief Scores (PRS) will be plotted against each timepoint up to the 1 hour timepoint, Total Pain Relief 0-1 hours (TOTPAR1) is the area under the curve. Each subjects TOTPAR1 will be expressed as a % of maxTOTPAR and compared to the slope of the change in pain intensity. The NRS will be used to assess the Pain Intensity, the NRS for pain is an 11-point scale (0-10) where a higher score indicates a greater amount of pain. PRS is a 5 point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?".
Relationship between speed of onset of pain relief and time to rescue medication over 0-60 minutes. | 0-1 hour
  To assess the relationship between speed of onset of pain relief and time to rescue medication by evaluating the association between the slope of the change in pain intensity over 0-60 minutes and time to rescue medication.

OTHER OUTCOMES:
Incidence of Treatment Emergent Adverse Events as assessed by patient response to questions and spontaneous reporting of TEAEs | 0-10 days
  Incidence of treatment emergent adverse events (TEAEs). Data listings will be provided for protocol specified safety data.
Vital signs measurements - Blood pressure in mm/Hg | 0-10 days
  Incidence of changes in vital sign measurements. Descriptive statistics will be provided at each scheduled time point for each treatment group. Changes from Baseline for vital signs will be calculated for each subject.
Vital signs measurements - Heart rate in beats per minute | 0-10 days
  Incidence of changes in vital sign measurements. Descriptive statistics will be provided at each scheduled time point for each treatment group. Changes from Baseline for vital signs will be calculated for each subject.
Vital signs measurements - Respiratory rate in breaths per minute | 0-10 days
  Incidence of changes in vital sign measurements. Descriptive statistics will be provided at each scheduled time point for each treatment group. Changes from Baseline for vital signs will be calculated for each subject
Vital signs measurements - Body Temperature in ºC | 0-10 days
  incidence of changes in vital sign measurements. Descriptive statistics will be provided at each scheduled time point for each treatment group. Changes from Baseline for vital signs will be calculated for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Davies NM. Clinical pharmacokinetics of ibuprofen. The first 30 years. Clin Pharmacokinet. 1998 Feb;34(2):101-54. doi: 10.2165/00003088-199834020-00002. PMID 9515184
- [Background] Cooper SA, Desjardins PJ, Turk DC, Dworkin RH, Katz NP, Kehlet H, Ballantyne JC, Burke LB, Carragee E, Cowan P, Croll S, Dionne RA, Farrar JT, Gilron I, Gordon DB, Iyengar S, Jay GW, Kalso EA, Kerns RD, McDermott MP, Raja SN, Rappaport BA, Rauschkolb C, Royal MA, Segerdahl M, Stauffer JW, Todd KH, Vanhove GF, Wallace MS, West C, White RE, Wu C. Research design considerations for single-dose analgesic clinical trials in acute pain: IMMPACT recommendations. Pain. 2016 Feb;157(2):288-301. doi: 10.1097/j.pain.0000000000000375. PMID 26683233
- [Background] Mehlisch DR, Sykes J. Ibuprofen blood plasma levels and onset of analgesia. Int J Clin Pract Suppl. 2013 Jan;(178):3-8. doi: 10.1111/ijcp.12053. PMID 23163542
- See also: Guidance for Industry Food-Effect Bioavailability and Fed Bioequivalence Studies — https://www.fda.gov/files/drugs/published/Food-Effect-Bioavailability-and-Fed-Bioequivalence-Studies.pdf#:~:text=This%20guidance%20provides%20recommendations%20to%20sponsors%20and%2For%20applicants,and%20fed%20BE%20studies%20should%20be%20performed.%202
- See also: Guideline on the clinical development of medicinal products intended for the treatment of pain — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-development-medicinal-products-intended-treatment-pain-first-version_en.pdf